CLINICAL TRIAL: NCT03557268
Title: Effects of Pubertal Blockade and Hormone Therapy on Cardiometabolic Risk Markers in Transgender Adolescents
Brief Title: Pubertal Blockade and Hormone Therapy in Transgender Youth
Acronym: PUBErTY
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 17-2328
Record Dates: First submitted 2018-05-08; First posted 2018-06-14 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Gender Identity; Gender Dysphoria; Gender Identity Disorder in Adolescence and Adulthood
MeSH Terms: conditions — Gender Dysphoria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Participants will have the options of banking plasma, serum, urine and stool for future research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- On a GnRHa: Half of subjects will be on a puberty blocker or gonadotropin-releasing hormone analogue
- Not on GnRHa: Half of subjects will NOT be on a puberty blocker or gonadotropin-releasing hormone analogue

SUMMARY:
This study will enroll female-to-male transgender youth who are and are not on a puberty blocker (gonadotropin-releasing hormone analogue) at baseline and 1 and 12 months after starting testosterone. The study will evaluate markers of cardiometabolic health including: insulin sensitivity, laboratory markers, vascular health, body composition, activity/fitness, mitochondrial function and the microbiome.

DETAILED DESCRIPTION:
There will be a total of 6 study visits: baseline A, baseline B, 1 month after starting testosterone (visit A and B) and 12 months after starting testosterone (visit A and B). No medications will be administered as a part of this study.

Visit A procedures: Physical Examination, Laboratory, and Oral Glucose Tolerance Test (OGTT) visit.

This will be conducted at Childrens Hospital Colorado (CHCO) Clinical & Translational Research Centers (CTRC) facilities. Physical examination will include vital signs, anthropometric measurements, and breast/pubic hair staging as applicable (some subjects may have already undergone mastectomy/chest masculinizing surgery) by the PI. Subjects will fast for 8 hours prior to blood draw. Fasting blood work will be obtained, followed by an oral glucose load (75g glucola). Blood glucose and insulin concentrations will be drawn at baseline and 30, 60, 90 and 120 minutes after glucola administration. Serum will be obtained at baseline and 2 hours post-OGTT and used for bile acid and lipid metabolomic profile. The following questionnaires will be administered: REDCap Health Questionnaire, PedsQLTM 4.0 generic core questionnaire, PROMIS Pediatric Anxiety Short Form, PROMIS Pediatric Depressive Symptoms Short Form, Insomnia Severity Index, Morningness and Eveningness Scale. Participants will be mailed or emailed the 3-day dietary log prior to the visit and return it at this visit. They will be given a stool microbiome collection kit and urine collection kit to return at visit B. The medical chart will be reviewed for relevant health information and medications.

Part B: Vascular Imaging, MR-based imaging and spectroscopy, Exercise Capacity and Dual-energy X-ray (DXA) visit.

This will be conducted at the University of Colorado Denver Energy Balance Core and UCD Brain Imaging Center. The participant will be fasting for a minimum of 4 hours prior to the beginning of the study visit. The investigators will perform the tests in the following order:

1. Participants will return stool microbiome and urine collection kit.
2. Vascular imaging: carotid artery stiffness and intimal medial thickness and brachial artery flow-mediated dilation
3. Magnetic Resonance (MR) based imaging and spectroscopy
4. Oxygen consumption (VO2) peak exercise test on a stationary bicycle.
5. Total body dual energy x-ray absorptiometry (DXA)
6. Participants will be provided with an accelerometer and actigraphy watch to wear for a period of 7 days to measure level of habitual physical activity and sleep, respectively. They will also be provided a handout with instructions and a sleep and activity diary to be filled out each day during the 7 days of wear.

ELIGIBILITY:
Inclusion Criteria:

* Identify as female-to-male
* Age 13-16 years at the time of enrollment
* If on a gonadotropin-releasing hormone analogue, > 6 months exposure
* Plan to start testosterone clinically in < 6 months.

Exclusion Criteria:

* Cognitive, psychiatric, or physical impairment resulting in inability to tolerate the study procedures
* Diabetes
* Antipsychotic medication
* Hypertension (resting BP ≥ 140/90 mm/Hg)
* Weight > 400 lbs (DXA and MRI limit)
* On estrogen and/or progesterone medications

Ages: 13 Years to 16 Years | Sex: Female
Age Groups: Child
Gender Based: Yes — Female-to-male transgender youth
Study Population: 16 female-to-male youth will be enrolled from 2 groups: 1) 8 female-to-male youth who have been on a gonadotropin-releasing hormone analogue for > 6 months; 2) 8 female-to-male (age-matched) youth who never received gonadotropin-releasing hormone analogue therapy.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Change in Insulin sensitivity | Baseline and 12 months after initiation of testosterone.
  Assessed by the Matsuda index, calculated from a 2-hour oral glucose tolerance test
Change in Vascular Health | Baseline and 12 months after initiation of testosterone.
  Brachial artery flow-mediated dilation

SECONDARY OUTCOMES:
Change in Mitochondrial function | Baseline and 12 months after initiation of testosterone.
  Hepatic mitochondrial function as assessed by 31Phosphorus- Magnetic Resonance Spectroscopy
Change in VO2 peak | Baseline and 12 months after initiation of testosterone.
  VO2 peak as measured on a bicycle ergometer
Change in Body composition | Baseline and 12 months after initiation of testosterone.
  as measured on a Dual-energy X-ray Absorptiometry (DXA) scan

CONTACTS AND LOCATIONS:
Overall Officials: Natalie J Nokoff, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided